CLINICAL TRIAL: NCT00685477
Title: Dose Response of Intravenous Sincalide (CCK-8) for Gallbladder Emptying
Brief Title: Dose Response of Intravenous Sincalide(CCK-8) for Gallbladder Emptying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Johns Hopkins University (Other); Penn State University (Other); Memorial Health University Medical Center (Other)
Responsible Party: Principal Investigator, Alan Maurer, Professor of Medicine, Temple University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: CCK-2008
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2016-12

CONDITIONS: Healthy
Keywords: CCK infusion; Gallbladder ejection fraction; Normal volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Experimental Sequence ABC (Active Comparator): CCK-8 0.02 mg/kg over 15 minutes, followed by CCK-8 0.02 mg/kg over 30 minutes, followed by CCK-8 0.02 mg/kg 60 minutes, with at least 2 days between each infusion
  Interventions: Drug: Experimental Sequence ABC
- Experimental Sequence ACB (Active Comparator): CCK-8 0.02 mg/kg over 15 minutes, followed by CCK-8 0.02 mg/kg over 60 minutes, followed by CCK-8 0.02 mg/kg 30 minutes, with at least 2 days between each infusion
  Interventions: Drug: Experimental Sequence ACB
- Experimental Sequence BAC (Active Comparator): CCK-8 0.02 mg/kg over 30 minutes, followed by CCK-8 0.02 mg/kg over 15 minutes, followed by CCK-8 0.02 mg/kg 60 minutes, with at least 2 days between each infusion
  Interventions: Drug: Experimental Sequence BAC
- Experimental Sequence BCA (Active Comparator): CCK-8 0.02 mg/kg over 30 minutes, followed by CCK-8 0.02 mg/kg over 60 minutes, followed by CCK-8 0.02 mg/kg 15 minutes, with at least 2 days between each infusion
  Interventions: Drug: Experimental Sequence BCA
- Experimental Sequence CAB (Active Comparator): CCK-8 0.02 mg/kg over 60 minutes, followed by CCK-8 0.02 mg/kg over 15 minutes, followed by CCK-8 0.02 mg/kg 30 minutes, with at least 2 days between each infusion
  Interventions: Drug: Experimental Sequence CAB
- Experimental Sequence CBA (Active Comparator): CCK-8 0.02 mg/kg over 60 minutes, followed by CCK-8 0.02 mg/kg over 30 minutes, followed by CCK-8 0.02 mg/kg 15 minutes, with at least 2 days between each infusion
  Interventions: Drug: Experimental Sequence CBA

INTERVENTIONS:
Drug: Experimental Sequence ABC — Drug will be given over 15 minutes, followed by infusion over 30 minutes, followed by infusion over 60 minutes
  Other Names: Sequence ABC
  Arms: Experimental Sequence ABC
Drug: Experimental Sequence ACB — Drug infused over 15 minutes, followed by infusion over 60 minutes, followed by infusion over 30 minutes
  Other Names: Sequence ACB
  Arms: Experimental Sequence ACB
Drug: Experimental Sequence BAC — Drug will be given over 30 min infusion, followed by 15 minute infusion, followed by 60 minute infusion
  Other Names: Sequence BAC
  Arms: Experimental Sequence BAC
Drug: Experimental Sequence BCA — Drug will be given over 30 min infusion, followed by 60 minute infusion, followed by 15 minute infusion
  Other Names: Sequence BCA
  Arms: Experimental Sequence BCA
Drug: Experimental Sequence CAB — Drug will be given over 60 min infusion, followed by 15 minute infusion, followed by 30 minute infusion
  Other Names: Sequence CAB
  Arms: Experimental Sequence CAB
Drug: Experimental Sequence CBA — Drug will be given over 60 min infusion, followed by 30 minute infusion, followed by 15 minute infusion
  Other Names: Sequence CBA
  Arms: Experimental Sequence CBA

SUMMARY:
This is a clinical research study to establish normal values for the infusion of a synthetic form of the hormone cholecystokinin(CCK-8) for gallbladder emptying. Cholecystokinin is released from the small bowel to stimulate the pancreas and gallbladder to help digest and absorb food. Some people have gallbladder problems and need to be tested with the synthetic cholecystokinin ( Kinevac®, Bracco Diagnostics, Inc.). The aim of this study is to find out how differing amounts and intravenous infusion times of CCK-8 affect gallbladder emptying. The findings in normal subjects will be used to establish normal values that can then be compared with patients with suspected gallbladder disease.

DETAILED DESCRIPTION:
This study enrolled 60 healthy volunteers from four institutions (Johns Hopkins University, Pennsylvania State University, Memorial Health University Medical Center, and Temple University. Subjects had to be healthy men or women 18-65 years old with no gastrointestinal disease as confirmed by initial screening using a modified Mayo Clinic Research Gastrointestinal Disease Screening Questionnaire, and normal results for CBC, metabolic profile, serum amylase and gallbladder ultrasonography. Women could not be enrolled if pregnant.

Subjects had 3 infusion studies at least 2 days apart within 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females between ages 18-65 years of age with no gastrointestinal disease as screened by the Mayo Clinic GI Disease Screening Questionnaire
2. Subjects with high probability for compliance and completion of the study
3. Normal liver function tests and amylase
4. Normal ultrasound of the gallbladder

Exclusion Criteria:

1. Prior GI surgery, excluding appendectomy
2. Surgery within the past 3 months
3. BMI > 35
4. Female of childbearing age who is not practicing birth control and/or is pregnant or lactating. (Confirm with urine pregnancy test)
5. Cardiovascular, endocrine, renal, gastrointestinal, or other chronic disease likely to affect motility. This includes diabetes, renal insufficiency, gastroesophageal reflux disease, gastroparesis, irritable bowel syndrome, prior peptic ulcer disease.
6. GI symptoms such as heartburn, chest pain, dysphagia, abdominal pain, nausea, vomiting, constipation, diarrhea.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan H Maurer, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Behar J, Corazziari E, Guelrud M, Hogan W, Sherman S, Toouli J. Functional gallbladder and sphincter of oddi disorders. Gastroenterology. 2006 Apr;130(5):1498-509. doi: 10.1053/j.gastro.2005.11.063. PMID 16678563
- [Result] Ziessman HA, Tulchinsky M, Lavely WC, Gaughan JP, Allen TW, Maru A, Parkman HP, Maurer AH. Sincalide-stimulated cholescintigraphy: a multicenter investigation to determine optimal infusion methodology and gallbladder ejection fraction normal values. J Nucl Med. 2010 Feb;51(2):277-81. doi: 10.2967/jnumed.109.069393. Epub 2010 Jan 15. PMID 20080900

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Sequence ABC: Drug given over 15 minutes infusion followed by infusion over 30 minutes, followed by infusion over 60 minutes
- Experimental Sequence ACB: Drug given over 15 minutes infusion followed by infusion over 60 minutes, followed by infusion over 30 minutes
- Experimental Sequence BAC: Drug given over 30 minutes infusion followed by infusion over 15 minutes, followed by infusion over 60 minutes
- Experimental Sequence BCA: Drug given over 30 minutes infusion followed by infusion over 60 minutes, followed by infusion over 15 minutes
- Experimental Sequence CAB: Drug given over 60 minutes infusion followed by infusion over 15 minutes, followed by infusion over 30 minutes
- Experimental Sequence CBA: Drug given over 60 minutes infusion followed by infusion over 30 minutes, followed by infusion over 15 minutes
Period: Overall Study
Arm/Group | Experimental Sequence ABC | Experimental Sequence ACB | Experimental Sequence BAC | Experimental Sequence BCA | Experimental Sequence CAB | Experimental Sequence CBA
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Each of the 60 subjects had 3 infusion studies at least 2 days apart.
Groups:
- All Study Participants: CCK-8 0.02 mg/kg over 15, 30 or 60 minutes: Drug will be given over infusions at different time periods. All participants received all treatments.
Arm/Group | All Study Participants
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (12)
Gender [Count of Participants; unit: Participants]
  Female | 32
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Coefficient of Variation (CV) for Gallbladder Ejection Fraction (GBEF) for Each Infusion Method
Description: The primary statistical endpoint was the CV as a measure of variability for the GBEF for each infusion method at the different intervals to determine which sincalide infusion method had the lowest variation. The CV is the SD divided by the mean and is expressed as a percentage and reflects the variability among the values. The infusion method having the lowest CV is considered best as it reflects the lowest variability of the values.
Time Frame: 15, 30, 45, and 60 minutes post drug infusion
Population: Some participants were excluded from analyses due to location testing procedures
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- 15min Infusion: Drug given over 15 minutes infusion
- 30 Min Infusion: Drug given over 30 minutes infusion
- 60 Min Infusion: Drug given over 60 minutes infusion
Arm/Group | 15min Infusion | 30 Min Infusion | 60 Min Infusion
Number analyzed (Participants) | 60 | 60 | 60
percentage
  15 min post infusion | 51.66 [43.79 to 63.01] | 62.75 [53.19 to 76.53] | 71.38 [60.52 to 87.08]
  30 min post infusion: number analyzed (Participants) | 45 | 60 | 60
  30 min post infusion | 40.46 [33.49 to 51.10] | 34.49 [29.23 to 42.06] | 35.81 [30.36 to 43.69]
  45 min post infusion: number analyzed (Participants) | 45 | 45 | 60
  45 min post infusion | 39.91 [33.05 to 50.42] | 31.30 [25.91 to 39.53] | 24.00 [20.35 to 29.28]
  60 min post infusion: number analyzed (Participants) | 45 | 45 | 60
  60 min post infusion | 35.21 [29.15 to 44.48] | 29.11 [24.10 to 36.77] | 18.55 [15.73 to 22.64]

2. Secondary Outcome: Gallbladder Ejection Fraction (GBEF) as a Percent for Each Infusion Method
Time Frame: 15, 30, 45 and 60 minutes post-infusion
Population: Some participants were excluded from analyses due to location testing procedures
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- 15 Minute Infusion: Drug given over 15 minutes
- 30 Minute Infusion: Drug given over 30 minutes
- 60 Minute Infusion: Drug given over 60 minutes
Arm/Group | 15 Minute Infusion | 30 Minute Infusion | 60 Minute Infusion
Number analyzed (Participants) | 60 | 60 | 60
percentage
  15 minutes post-infusion | 57 (29) | 44 (28) | 34 (24)
  30 minutes post-infusion: number analyzed (Participants) | 45 | 60 | 60
  30 minutes post-infusion | 67 (27) | 71 (24) | 64 (23)
  45 minutes post-infusion: number analyzed (Participants) | 45 | 45 | 60
  45 minutes post-infusion | 66 (26) | 73 (23) | 78 (19)
  60 minutes post-infusion: number analyzed (Participants) | 45 | 45 | 60
  60 minutes post-infusion | 68 (24) | 74 (21) | 84 (16)

ADVERSE EVENTS:
Time Frame: 15 min, 30 min, 45 min, and 60 min post-infusion
Groups:
- All Study Participants: Drug given over 15 minute infusion to look at lowest coefficient of variation in infusion, followed by infusion over 30 minutes, followed by infusion over 60 minutes
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No